CLINICAL TRIAL: NCT06169345
Title: The Long-term Clinical Course of Moderate Tricuspid Regurgitation
Brief Title: The Long-term Course of Moderate Tricuspid Regurgitation
Acronym: LOCOMOTRI
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Agricola Eustachio, Director of Cardiovascular Imaging Department, IRCCS San Raffaele
Other Study IDs: LOCOMOTRI STUDY
Record Dates: First submitted 2023-09-26; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Tricuspid Regurgitation; Heart Failure; Echocardiography
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Echocardiographic evaluation — Echocardiographic follow-up

SUMMARY:
To evaluate the long-term clinical outcome of a cohort of patients suffering from moderate tricuspid regurgitation (TR), regardless of its etiology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an echocardiographic diagnosis of moderate TR
2. Patients with echocardiographic and clinical follow-up information available at least 6-months after moderateTR diagnosis.

Exclusion Criteria:

1. Absence of an appropriate clinical and echocardiographic follow-up
2. A history of previous TV intervention (either surgical or percutaneous)
3. The presence of concomitant TV stenosis
4. Congenital heart disease
5. Left ventricular assist devices

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with an echocardiographic diagnosis of moderate tricuspid regurgitation at our center between 2010 and 2019
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
All-cause death | through study completion, an average of 2 years
  Time from diagnosis to all-cause death

SECONDARY OUTCOMES:
Cardiovascular (CV) mortality | through study completion, an average of 2 years
  The occurrence of cardiovascular (CV) mortality (defined as death due to advanced heart failure, coronary ischemic heart disease, sudden cardiac death or due to stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No